CLINICAL TRIAL: NCT00463372
Title: A Phase I, Investigator And Subject-Blind (Sponsor Unblinded), Placebo-Controlled Dose Escalation Study To Evaluate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Pf-02545920 After Multiple Oral Dose Administration In Subjects With Stable Schizophrenia
Brief Title: Study Investigating the Safety and Tolerability of Multiple Doses of PF-02545920 in Subjects With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A8241002
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2007-09

CONDITIONS: Schizophrenia; Schizo-affective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — 2-((4-(1-methyl-4-pyridin-4-yl-1H-pyrazol-3-yl)phenoxy)methyl)quinoline

INTERVENTIONS:
Drug: PF-02545920

SUMMARY:
To evaluate the safety and tolerability of multiple doses of PF-02545920 subjects with schizophrenia or schizo-affective disorder who are currently clinically stable and to evaluate the serum and urine pharmacokinetics of PF-02545920 and the N-desmethyl metabolite, PF-01001252, after multiple doses of PF-02545920 administered orally.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with DSM-IV diagnosis of schizophrenia or schizo-affective disorder for whom antipsychotic monotherapy is indicated.
* Subjects must be free from an acute exacerbation of psychosis for at least 3 months prior to screening.
* Current Clinical Global Impression (CGI) of Severity of Illness score ≤ 3.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Evidence or history of a primary DSM-IV axis I diagnosis other than schizophrenia or schizoaffective disorder.
* Any condition possibly affecting drug absorption (e.g., gastrectomy).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40
Dates: Start 2006-10; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Safety endpoints: physical and neurological examination, adverse event reports, clinical laboratory tests, vital signs, and 12-lead ECGs throughout the conduct of the study.
Pharmacokinetic endpoints: Primary: AUCtau, Tmax and Cmax of PF-02545920 and PF-01001252 on Days 1 and 13.

SECONDARY OUTCOMES:
Secondary efficacy endpoints include: PANSS, CGI-S, CGI-I, CDSS, CNSVS VS-M cognitive battery, ESRS-A and SSS change from baseline to day 12.
Secondary PK endpoints include AUClast, t1/2, Cavg, Cmax/Cmin ratio on Day 13, and urinary excretion parameters (renal clearance and amount excreted over the dosing interval) of PF-02545920 and PF-01001252 as data permit.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, George, South Africa

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8241002&StudyName=Study+investigating+the+safety+and+tolerability+of+multiple+doses+of+PF%2D02545920+in+subjects+with+schizophrenia